CLINICAL TRIAL: NCT07071103
Title: Efficacy and Safety of Combining Intestinal Low Dose Radiotherapy and PD-1/PD-L1 Inhibitors for Metastatic Malignant Solid Tumors After Acquired Resistance to Anti-PD1/PD-L1 Treatment
Brief Title: Intestinal Low Dose Radiotherapy Combined With Immunotherapy in Immune-resistant Metastatic Malignant Solid Tumors
Acronym: ILDR-02
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chuangzhen Chen (Other)
Responsible Party: Sponsor-Investigator, Chuangzhen Chen, Director, Shantou University Medical College
Organization: Shantou University Medical College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUMC-ILDR02
Record Dates: First submitted 2025-07-09; First posted 2025-07-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Radiotherapy; Metastatic Solid Cancers; Immune Checkpoint Blockade; Esophageal Neoplasms Malignant; Lung Neoplasm Malignant; Drug Resistance
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lung cancer arm (Experimental): This arm includes patients with metastatic non-small cell lung cancer (NSCLC) or small cell lung cancer (SCLC) who have progressed after previous immune checkpoint blockades (ICBs) administration, and the intervention involves 1Gy/1F ILDR plus PD-1/PD-L1 inhibitors.
  Interventions: Radiation: Low-dose radiotherapy to the intestine (ILDR); Drug: PD-1/PD-L1 monoclonal antibodies
- Esophageal cancer group (Experimental): This arm includes patients with metastatic esophageal cancer (including squamous cell carcinoma or adenocarcinoma) who have progressed after previous ICB administration, and the intervention involves 1Gy/1F ILDR plus PD-1/PD-L1 inhibitors.
  Interventions: Radiation: Low-dose radiotherapy to the intestine (ILDR); Drug: PD-1/PD-L1 monoclonal antibodies
- Other solid tumor group (Experimental): This arm includes patients with other malignant solid tumors except lung cancer and esophageal cancer who have progressed after previous ICB administration, and the intervention involves 1Gy/1F ILDR plus PD-1/PD-L1 inhibitors.
  Interventions: Radiation: Low-dose radiotherapy to the intestine (ILDR); Drug: PD-1/PD-L1 monoclonal antibodies

INTERVENTIONS:
Radiation: Low-dose radiotherapy to the intestine (ILDR) — A single total dose of 1 Gy irradiation targeting the jejunum and ileum. Primary tumor or metastatic lesions that are within the irradiation field are irradiated concurrently.
Drug: PD-1/PD-L1 monoclonal antibodies — Pre-progression immunotherapy regimen continues or switches to an alternative PD-1/PD-L1 monoclonal antibody according to clinical guidelines.PD-1/PD-L1 monoclonal antibody will be given 1 day after ILDR at a 3-week interval.

SUMMARY:
Preclinical and clinical evidence suggests that intestinal low-dose radiotherapy (ILDR) may enhance antitumor immune responses by modulating the gut microenvironment, thereby improving the efficacy of immune checkpoint inhibitors (ICBs) in refractory solid tumors. Based on these findings, the investigators initiate a multicohort phase II clinical trial to evaluate the clinical benefit and safety of ILDR combined with PD-1/PD-L1 monoclonal antibody therapy in patients with metastatic solid tumors resistant to prior ICB treatment.

In this study, patients are stratified into three parallel cohorts by tumor type (lung cancer, esophageal cancer, and other solid tumors), with 16 patients per cohort (48 in total, including subjects enrolled from the ILDR-01 study). Eligible participants includes patients with advanced metastatic solid tumors progressing after monotherapy or combination ICB treatment, meeting criteria of ECOG performance status 0-2, life expectancy ≥3 months, and have at least one measurable lesion. Exclusion criteria encompasses prior pelvic radiotherapy, ongoing infections, major organ dysfunction, or concurrent antitumor therapies.

The primary endpoints includes objective response rate (ORR), disease control rate (DCR), progression-free survival after ILDR (PFS2), and the incidence of abscopal effects. Secondary endpoints includes overall survival (OS), treatment safety, α/β diversity changes in gut microbiota, peripheral blood immune cell subset dynamics, and tumor immune microenvironment remodeling characteristics. All patients receives a 1 Gy jejunoileal radiotherapy followed by PD-1/PD-L1 monoclonal antibody administration (in accordance to prior protocols or guidelines) within 24 hours, with maintenance therapy up to 2 years. Therapeutic efficacy is assessed via RECIST v1.1, while therapeutic toxicity is assessed according to CTCAE v5.0.

Paired pre- and post-treatment samples (including wumor tissue, stool, peripheral blood etc.) are collected for metagenomic sequencing, metabolomic analysis, and multi-omics integrative modeling to systematically elucidate the regulation mechanism of gut microbiota-metabolite-immune axis mediated by ILDR. This approach aims to provide theoretical foundations for optimizing treatment strategies in immunotherapy-resistant tumors and identify biomarkers that potentially associated with therapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, ≤80 years, regardless of gender.
* ECOG level 0-2.
* Expected life span>3 months.
* At least one accessible and measurable lesion should be selected as the target lesion for observation according to RECIST criteria.
* Patients with metastatic solid tumors (of any histology) without standard therapy options, who have previously received immunotherapy, immunotherapy combined with chemotherapy, or immunotherapy combined with anti-angiogenesis treatment and have shown disease progression.
* Patients should not be considered eligible for surgical treatment.
* Patients with brain metastases that are assessed as clinically stable after treatment through repeated CT and/or MRI scans are eligible.
* Patients have complete clinical and pathological information.
* Patients should not be borthered by any psychological, family, social or geographical conditions that may hinder compliance with the research protocol.
* Patients should be able to understand the informed consent form, voluntarily participate, and sign the informed consent form.
* Other indicators accord with the general inclusion criteria for clinical trials.

Exclusion Criteria:

* Patients with contraindications to radiation therapy and immunotherapy.
* Previous occurrence of unacceptable immune related toxic side effects (immune myocarditis, pneumonia, etc.).
* Patients who were assessed as hyperprogressive disease (HPD).
* Patients who have received pelvic and abdominal radiation therapy within 6 months prior to enrollment.
* The adverse reactions from prior treatment have not yet recovered to a CTCAE5.0 rating of ≤ 1 (excluding toxicity that has been determined to be risk-free, such as fatigue or hair loss).
* Patients with active uncontrolled systemic bacterial, viral, or fungal infections despite optimal treatment.
* Significant liver or kidney dysfunction (i.e., laboratory values >3 times the upper limit of normal).
* Active hepatitis B, hepatitis C, HIV, or syphilis.
* Brain disorders, symptomatic central nervous system (CNS) or meningeal metastases, or impaired cognitive function.
* Hypersensitivity to any drug included in the trial.
* Drug and/or alcohol abuse.
* Pregnant or breastfeeding women.
* Concurrent participation in another therapeutic clinical trial.
* Poorly controlled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within ≤14 days after intervention).
* Major surgery within 30 days.
* Use of antibiotics, antifungals, antivirals, antiparasitics, or probiotics within 4 weeks before enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 6, 12, 24 weeks after ILDR initiation.
  Proportion of patients achieving complete response (CR) or partial response (PR) (sustained ≥4 weeks) per RECIST v1.1.
Disease Control Rate（DCR） | 6, 12, 24 weeks after ILDR initiation.
  Proportion of patients with CR, PR, or stable disease (SD) per RECIST v1.1.
Progression Free Survival while Receiving ILDR combined Therapy (PFS2) | 6, 12, 24 weeks after ILDR initiation.
  Time from ILDR treatment to second documented disease progression (assessed by investigator via PSA, imaging, symptom, or the combinations) or death from any cause.
Incidence of Abscopal Effect | 6, 12, 24 weeks after ILDR initiation.
  Proportion of patients demonstrating tumor response in one or more non-irradiated lesions.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24, 48 weeks after radiotherapy initiation.
  Time from ILDR treatment initiation to death from any cause.
Cancer-Specific Survival (CSS) | 24, 48 weeks after radiotherapy initiation.
  Time from ILDR treatment initiation to death due to cancer.
Adverse Events | 12, 24, 48 weeks after radiotherapy initiation
  Proportion of patients with treatment-related adverse events as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Peripheral Blood Analyses | Before the first ILDR, 3-7 days after ILDR initiation, before each subsequent administration of the PD-1/PD-L1 blockade.
  Peripheral blood analysis includes immune profiling, transcriptomics, immune receptor repertoire, metabolomics, and cytokine analysis
Tissue Analyses | Before the first ILDR, 3 weeks after the last ILDR or before the next PD-1/PD-L1 blockade administration.
  Tissue analyses includes transcriptomics, immune receptor repertoire, and immunohistochemistry.
Fecal Analyses | Before the first ILDR, 3-7 days after each ILDR, after each subsequent PD-1/PD-L1 blockade administration.
  Fecal analyses include fecal metagenomics and fecal metabolomics.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No